CLINICAL TRIAL: NCT06465407
Title: Effect of Collagen Protein Versus Placebo on Indirect Markers of Musculotendinous Unit Recovery Following Eccentric Plantar Flexor Exercise
Brief Title: Collagen Protein Versus Placebo on Muscle Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Ecaterina Vasenina, Graduate Research Associate, University of Central Florida
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: UCFlorida1
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Anthropometrics: Height and Weight; Isometric Standing and Seated Plantarflexion; Calf Muscle Thickness; Achilles Tendon Length and Thickness; Myotonography of the Calf Musculature and Achilles Tendon; Pain Pressure Threshold of the Calf; Pain Scale; Endurance Calf Test; Dietary Analysis
MeSH Terms: conditions — Body Weight | interventions — Collagen; maltodextrin

STUDY DESIGN:
Intervention Model Description: This is a single blind repeated measures study design. There will be an intervention group and a control group. Intervention group is sub-divided into those who receive collagen (n=12) and those who receive placebo (n=12). The intervention group will perform every assessment including a standardized exercise routine focused on eccentric movements. Control group (n=12) will receive no supplement. Control group participants will do all the assessments that the intervention participants are performing, except for the standardized exercise routine focused on the eccentric movements. Randomization will be performed via www.randomizer.org website.
Who Masked: Participant
Masking Description: Single blind repeated measures design. Participants will be blinded to the intervention while research team will not be blinded and will be mixing supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen (Experimental): Collagen supplementation group will have 12 participants. They will perform various physical assessments that include pain scale, pain pressure threshold assessment, body composition, calf circumference measurements, muscle thickness measurements, Achilles tendon length and thickness measurements, myotonography of the calf, isometric force assessments during standing and seated plantarflexion positions, a heel raise test, and a standardized exercise routine focused on eccentric movements, targeting a leg chosen at random. Additionally, they will consume a daily dose of two 30-g amount of collagen peptides derived from bovine hide (commercially available as Vital Proteins or Peptan).
  Interventions: Dietary Supplement: Collagen
- Placebo (Placebo Comparator): Placebo supplementation group will have 12 participants. They will perform various physical assessments that include pain scale, pain pressure threshold assessment, body composition, calf circumference measurements, muscle thickness measurements, Achilles tendon length and thickness measurements, myotonography of the calf, isometric force assessments during standing and seated plantarflexion positions, a heel raise test, and a standardized exercise routine focused on eccentric movements, targeting a leg chosen at random. Additionally, they will consume a daily dose of placebo (two 30 g of pure maltodextrin with no amino acids) mixed in 300 ml of orange Gatorade zero.
  Interventions: Dietary Supplement: Maltodextrin
- Control (No Intervention): Control group (n=12) will receive no supplement. Control group participants will do all the assessments that the intervention participants are performing, except for the standardized exercise routine focused on the eccentric movements. Randomization will be performed via www.randomizer.org website.

INTERVENTIONS:
Dietary Supplement: Collagen — Participants will consume two 30-g amount of collagen peptides derived from bovine hide (commercially available as Vital Proteins or Peptan) mixed in 300 ml of orange gatorade zero.
  Arms: Collagen
Dietary Supplement: Maltodextrin — Participants will consume two 30-g amount of pure maltodextrin mixed in 300 ml of orange gatorade zero.
  Arms: Placebo

SUMMARY:
This study is focused on exploring the gap in the literature by comparing the effects of collagen protein versus placebo supplementation on the musculotendinous unit following muscle damaging protocol. Thus, the purpose of this study is to identify and compare the effect of collagen protein versus placebo supplementation on indirect markers of musculotendinous unit recovery following eccentric calf exercises.

DETAILED DESCRIPTION:
Various physical assessments that include pain scale, pain pressure threshold assessment, body composition, calf circumference measurements, muscle thickness measurements, Achilles tendon length and thickness measurements, myotonography of the calf, isometric force assessments during standing and seated plantarflexion positions, a heel raise test, and a standardized exercise routine focused on eccentric movements, targeting a leg chosen at random. Additionally, will consume a daily dose of two 30-g amount of collagen peptides derived from bovine hide (commercially available as Vital Proteins or Peptan) or placebo (30 g of pure maltodextrin with no amino acids) mixed in 300 ml of orange Gatorade zero.

Gatorade zero, maltodextrin, and collagen is going to be stored in the locked cabinet in the lab. Research team will mix the supplement (placebo or maltodextrin) with Gatorade zero in a non-clear bottle and will administer it to the participants on-site.

ELIGIBILITY:
Inclusion Criteria:

* Males between the ages of 18-30 years old
* Determined to be healthy by PAR-Q+ and the HHQ

Exclusion Criteria:

* Untrained (no resistance training in the past 3 months)
* Any response of "yes" on the PAR-Q+; exclusion criteria noted on the HHQ
* Allergy to bovine collagen or maltodextrin

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males between the ages of 18-30 years old
Enrollment: 36 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Calf muscle thickness | 5 days
  Portable B-mode Ultrasound (GE Logiq e BT12, GE Healthcare, Milwaukee, WI, USA) and a multi-frequency linear- array probe (12 L-RS, 5-13 MHz, 38.4-mm field of view, GE Healthcare, Milwaukee, WI, USA) will be used to determine changes in muscle thickness of the randomized leg. The distance between the medial point of the knee joint space and the central point of the medial malleolus will be measured at 70% and ultrasound gel will be placed on this location prior to measurement. The highest and mean values of 3-5 measurements will be recorded for each assessment. All measurements will be done on one randomized leg.

SECONDARY OUTCOMES:
Achilles tendon thickness. | 5 days
  Achilles tendon will be scanned using a B-mode US imaging device (GE Logiq e, GE Healthcare,Wauwatosa, WI, USA) and a multi-frequency linear-array probe (12 L-RS, 5-13 MHz, 38.4-mm field of view; GE Healthcare). The same researcher will perform the assessments. All ultrasound imaging analyses will be performed using Image-J software 1.8.0 (National Institute of Health, Bethesda, MD, USA). Achilles tendon length will be determined using the segmented line function between calcaneal notch and muscle-tendon junction along the midline of the Achilles tendon. Additionally, sagittal images of the Achilles tendon will be collected with the ankle passively dorsiflexed to approximately 90 degrees. Tendon thickness will be measured at reference point of 2 cm proximal to the superior aspect of the calcaneus.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided